CLINICAL TRIAL: NCT06828315
Title: Foot Reflexology as an Adjunctive Therapy in Migraine Management: A Randomized Controlled Trial on Pain, Fatigue, and Quality of Life
Brief Title: the Effect of Reflexology in Migraine Patients
Acronym: migraine
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Cihat Demirel, Assistant Professor, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: migraine
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Reflexology; Migraine; Pain; Fatigue; Quality of Life
MeSH Terms: conditions — Migraine Disorders; Pain; Fatigue | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): reflexology was applied to the experimental group
  Interventions: Other: Reflexology
- control group (No Intervention): reflexology was not applied to the control group

INTERVENTIONS:
Other: Reflexology — Reflexology is a practice based on the fact that the organs in the body are connected to the reflex areas in the hands and feet.
  Arms: experimental group

SUMMARY:
The aim of this randomised controlled trial was to evaluate the effect of foot reflexology on pain intensity, fatigue and quality of life in migraine patients.

The main questions it aims to answer are:

Is foot reflexology effective in reducing pain intensity in migraine patients? Is foot reflexology effective in reducing the fatigue level of migraine patients? Is foot reflexology effective in improving the quality of life of migraine patients? Comparison group: The researchers will evaluate the effects of foot reflexology by comparing the group receiving reflexology intervention with the control group receiving only routine treatment.

Participants were selected according to the following criteria:

Intervention group: Individuals diagnosed with migraine will receive foot reflexology twice a week for a total of 10 sessions.

Control group: No additional intervention will be applied to this group, only their routine treatment and medical follow-up will continue.

Both groups will be evaluated at the beginning and at the end of the study with the Patient Information Form, Migraine 24-Hour Quality of Life Scale (QoLQS), Visual Analogue Scale (VAS) and Fatigue Severity Scale (FSS). After the completion of the study, reflexology will be applied to patients in the control group who are willing to receive reflexology.

ELIGIBILITY:
Inclusion Criteria:

1. Being between the ages of 18-60 (to conduct the study with adult individuals and to minimise the effect of age-related variables)
2. Being diagnosed with migraine
3. Having experienced at least 2 migraine attacks in the last 6 months (to ensure a homogenous group among patients with more chronic or episodic migraine)
4. Migraine with a severity of 4 or more with VAS (Visual Analogue Scale) (To prevent mild headaches from affecting the study)
5. Having experienced at least 2 migraine attacks in the last 6 months (to ensure a homogenous group among patients with more chronic or episodic migraine)
6. To participate and continue to work as a volunteer

Exclusion Criteria:

1. For female participants: Being pregnant or breastfeeding (as hormone changes may change the effect of migraine and reflexology)
2. Having another chronic neurological disease (epilepsy, MS, Parkinson's, etc.) (to avoid the effect of symptoms that may be confused with migraine)
3. Being treated with another alternative medicine method (acupuncture, biofeedback, etc.) at the same time (to measure the independent effect of reflexology)
4. Regular use of Botox, nerve blockade or invasive treatment for migraine in the last 3 months (to reduce the influence of external factors on migraine severity)
5. Severe psychiatric disorders (schizophrenia, bipolar disorder, etc.) or a history of severe depression/anxiety (to isolate the effect of stress and psychological factors on reflexology)
6. No previous serious side effects or intolerance to reflexology (important for safety)
7. Diabetic neuropathy, severe peripheral neuropathy or severe dermatological disorders (infection, open wound, etc.) in the foot area (as it may affect the applicability of reflexology)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2025-02-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | At the end of the 5-week intervention
  The Visual Analog Scale (VAS) will be used to assess the change in pain intensity before and after the intervention. Participants will rate their migraine pain on a 10 cm scale, where 0 represents "no pain" and 10 represents "worst pain imaginable."
Fatigue Severity Scale (FSS) | At the end of the 5-week intervention
  The Fatigue Severity Scale (FSS) will be used to evaluate changes in participants' fatigue levels. The FSS consists of nine items scored from 1 to 7, with higher scores indicating greater fatigue severity.
24-Hour Migraine-Specific Quality of Life Questionnaire (24 h MQoLQ) | At the end of the 5-week intervention
  24-Hour Migraine-Specific Quality of Life Questionnaire (24 h MQoLQ) will assess changes in migraine-specific quality of life. It includes five subscales: Migraine Symptoms, Emotions and Concerns, Work Functionality, Social Functionality, and Energy/Vitality. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Cihat Demirel, Principal Investigator — Muş Alparslan University
Locations (1):
- Muş Alparslan University, Muş, Turkey (Türkiye)